CLINICAL TRIAL: NCT01929369
Title: Pilot Study of IVUS Imaging During Endovascular Interventions of Failing Hemodialysis Access Grafts
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Ross Pilot
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: THROMBOSED AV GRAFTS
Keywords: ESRD; CKD; AV GRAFTS; THROMBOSED AV GRAFTS
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CONTROL GROUP: Control group: index intervention guided by DSA; IVUS post-intervention only (50 patients)
- TEST GROUP: Test group: index intervention guided by IVUS + DSA (50 patients

SUMMARY:
This pilot study will provide data to aid in the planning of a follow-up multi-center randomized, controlled trial (RCT). As such, the sample size for this pilot is not driven by formal statistical hypothesis testing. Rather, the sample size of 100 patients (50 per arm) was derived in consultation with the study PI and Co-PI who are experts in vascular surgery, and in particular, the field of hemodialysis access interventions. The results of this pilot study will provide the data that is necessary for generation of specific hypotheses that can then be formally tested in the follow-up RCT

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be > 18 and < 85 years of age
2. Patient or legally authorized representative must be willing to participate and able to understand, read, and sign the informed consent document before the planned procedure
3. Eligible for de-clot procedure or evaluation of slow flow for a failing hemodialysis graft that previously provided access for at least 1 successful hemodialysis session

Exclusion Criteria:

1. Patient or legally authorized representative cannot or will not provide written informed consent
2. Known metal allergy precluding endovascular stent implantation
3. Known reaction or sensitivity to iodinated contrast that cannot be pretreated
4. Patients who are pregnant or lactating
5. Patients with scheduled kidney transplant within the next 6 months
6. Patients scheduled to switch to peritoneal dialysis within the next 6 months
7. Patients with life expectancy of less than 6 months
8. Participation in any other clinical research study that would interfere with the patient's participation in this study
9. Any concurrent disease or condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD PATIENTS WITH THROMBOSED AV GRAFTS
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Re-Intervention Control vs. Test | 6 months
  Difference in time (measured in days) to AV graft failure after index intervention guided by DSA in the absence (control group) or presence of IVUS guidance (test group), assessed through 6 months post-index procedure
Define IVUS workflow | Day 0
  Define IVUS workflow for AV graft evaluation during interventions for access site failure
Evaluate ability of IVUS in AV Grafts | Day 0
  Evaluate the ability of IVUS to identify targets for therapy in poorly functioning AV grafts that are not identified by DSA

SECONDARY OUTCOMES:
IVUS vs DSA alone- Decision making | Day 0
  Percentage of time IVUS changes decision making during the index procedure (test group)
% patients requiring re-intervention | 3 months and 6 months
  Percentage of patients with graft failure or need for reintervention at 3 months and 6 months (c0ntrol and test)
Assess CHROMOFLO in AV grafts | Day 0
  Assess the ability of ChromaFlo® to identify residual thrombus in the hemodialysis access circuit

CONTACTS AND LOCATIONS:
Overall Officials: John Ross, MD, Principal Investigator — Regional Medical Center
Locations (1):
- Regional Medical Center, Orangeburg, South Carolina, United States